CLINICAL TRIAL: NCT02765685
Title: Randomized Controlled Trial in Internal Compartment Knee Osteoarthritis: ODRA Made-to-measure Hinged Knee Brace Versus Usual Care.
Brief Title: Internal Compartment Knee Osteoarthritis: ODRA (Orthosis Distraction and Rotation for osteoArthritis) Made-to-measure Hinged Knee Brace Versus Usual Care.
Acronym: ERGONOMIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ORNETTI 2013
Record Dates: First submitted 2016-04-29; First posted 2016-05-09 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (2):
- ODRA (Experimental)
  Interventions: Device: brace ODRA (PROTEOR company); Other: Usual care
- usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Device: brace ODRA (PROTEOR company) — Port of the orthosis ODRA during day during 12 months, Complement to their usual care. The subjects will have for instruction to wear the brace a minimum of 6 hours a day, 5 days a week, And to remove it during the rest periods in lengthened position.
  Arms: ODRA
Other: Usual care — The patients will benefit only from the coverage proposed usually, by their regular doctor and according to the notices of the medical and paramedical specialists taking care of this pathology (physiotherapists, orthopaedic osteopaths, sports medicine physician, surgeon, rheumatologists, rehabilitative doctors, etc.). In the absence of recommendations on the modalities of coverage of the gonarthrose and in front of diverse clinical habits, the "usual" said coverage can be at the same time medicinal (anti-inflammatory, painkilling, …), non-medicinal (physiotherapy, port of an orthosis, …), even surgical, according to the influencers.

SUMMARY:
This is a biomedical study on a medical device. 120 patients will participate in this study and will be split into 2 groups:

* 60 patients in the "usual care" group: these patients will receive the usual care proposed by their doctor for 12 months.
* 60 patients in the "ODRA" group: these patients will wear the ODRA brace for 12 months in addition to their usual care. They will be instructed to wear the brace for at least 6 hours per day, 5 days per week and to take it off during rest periods when lying down.

The distribution of patients in the groups will be randomized. For this study, patients will be followed for 12 months, spread over 3 visits: inclusion visit, follow-up visit at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Knee osteoarthritis (defined according to American College of Reumatology criteria):

  * radiological stage II, III or IV according to the Kellgren and Lawrence (KL) classification documented by a radiological examination in the previous 12 months.
  * Predominantly affecting the internal compartment (internal KL stage greater than external KL stage) and symptomatic with a Pain Visual Analogue Scale > 40/100 on the target side (side with the most symptomatic disease)
* Patients who have provided written consent
* Patients able to understand simple instructions, to read, write, and to give informed consent
* Patients with national health insurance cover

Exclusion Criteria:

* Severe venous insufficiency in the lower limbs
* History of deep venous thrombosis in the lower limbs
* Inflammatory flare of knee osteoarthritis (synovial effusion) on the target side
* Person over 18 under guardianship or unable to provide consent
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pain measured using a VAS (visual analogue scale) by the patient | 12 months

SECONDARY OUTCOMES:
Ratio differential cost-utility | 12 months
Evolution of pain measured by VAS in the form of a self-questionnaire | 6 months
Evolution of the Function score- Everyday life of the KOOS (Knee injury and osteoarthritis outcome score) self-questionnaire | 12 months
Evolution of quality of life measured by the AMIQUAL self-questionnaire | 12 months
Evolution de overall disease activity measured by VAS | 12 months
Consumption of care relative to the knee osteoarthritis | 12 months
  Surgical operation, injectable medicinal treatments and anti-osteoarthritic of slow action, care of Support
Local or general adverse effects | 12 months
Compliance with wearing the brace | 12 months
  Average number of hours of port of the brace a day, the average number of days of port of the brace a week. The possible motives for non-observance will be brought together.
  The patient will be considered compliant if he carries his brace at least 15 hours a week on average.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France